CLINICAL TRIAL: NCT04729829
Title: A Randomised Controlled Trial to Test the Effects of Fish Aggregating Devices and SBC Activities Promoting Fish Consumption in Timor-Leste
Brief Title: Fish Consumption and Dietary Diversity in Timor-Leste
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: WorldFish (Other)
Collaborators: Mercy Corps (Other)
Responsible Party: Principal Investigator, Alex Tilley, Principle Investigator, WorldFish
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: FSSP2_RCT1
Record Dates: First submitted 2021-01-25; First posted 2021-01-29 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Dietary Deficiency
Keywords: fish; fish aggregating device; malnutrition; micronutrient deficiency; fisheries
MeSH Terms: conditions — Malnutrition | interventions — Flavin-Adenine Dinucleotide

STUDY DESIGN:
Intervention Model Description: The main treatment variable is a dummy variable that indicates to which of the four treatment arms a village was assigned. Our primary model is an unadjusted model. However, if we find that after unmasking, there are variables in the dataset that appear different by treatment arm, we may consider adjusting for confounders in the model.
  We will first estimate a parsimonious model with only the treatment dummies and the municipality fixed effects. Then we will control for additional baseline covariates. The control group is the no-FAD and no-SBC group. Intent to treat (ITT) will be estimated separately for midline and end line subsamples. However, we will compare the magnitude of impacts at midline and endline.
Who Masked: Outcomes Assessor
Masking Description: Partially masked. Participation is randomised to the community level. Participants will be aware they are participating in a project/study, but not the particular study design or which treatment arm they are assigned to. Statistical analysts will be masked until the analysis is complete.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- FAD + SBC (Active Comparator): Community will be exposed to increased availability of fish from a fish aggregating device and will receive information and messaging as part of a social and behaviour change communication about consuming fish.
  Interventions: Behavioral: Social and behaviour change communication; Other: Fish aggregating device
- FAD only (Active Comparator): Community will be exposed to increased availability of fish from a fish aggregating device only
  Interventions: Other: Fish aggregating device
- SBC only (Active Comparator): Community will receive information and messaging as part of a social and behaviour change communication about consuming fish.
  Interventions: Behavioral: Social and behaviour change communication
- Control (No Intervention): Control (No FAD or SBC)

INTERVENTIONS:
Behavioral: Social and behaviour change communication — Each SBC treatment community will receive nutrition content and learning through savings groups. The group members will participate in skill-building activities that promote five key behaviours about fish nutrition and household decision making on fish consumption as part of facilitated discussions, interactive learning sessions, and a video-based facilitated dialogue. Increased fish consumption through SBC mass attendance events through marketing of fish vendors, interactive learning, and edu-tainment competitions promoting fish consumption. SBC will raise awareness of the benefits of eating fish as part of a balanced diet, with a particular focus on pregnant and lactating mothers, and children under 5 years of age.
  Arms: FAD + SBC; SBC only
Other: Fish aggregating device — This is a moored line attached to buoys in coastal waters that attracts oceanic fish to it, to make it easier for small-scale fishers to catch them using their existing gear and boats. This FAD will work to increase the catch rate and hence, the availability of fish for sale in upland community markets.
  Other Names: FAD
  Arms: FAD + SBC; FAD only

SUMMARY:
A one-year, cluster-randomized, partially masked, controlled trial to test and compare the effects of fish aggregating devices and social and behaviour change communication on the frequency and volume of household fish consumption in upland areas of Timor-Leste.

DETAILED DESCRIPTION:
This trial is a one-year, cluster-randomized, partially masked, controlled trial among families living in rural, inland Timor-Leste. This trial aims to test and compare the effects of two treatments, alone and in combination, on the frequency and volume of household fish consumption in upland areas as a proxy for improved dietary diversity and micronutrient intake. Treatment 1 is the installation of nearshore, moored fish aggregating devices (FADs) to improve catch rates with existing fishing gears. Treatment 2 is social and behaviour change (SBC) activities to promote fish consumption. Villages in inland communities will be randomized to receive treatment 1, treatment 2, both treatments, or neither treatment. Some households with one child under five will be recruited, and data will be collected at baseline (prior to the rollout of the treatments) and endline. Our study will determine the impact of an improved supply of fish, along with nutrition-oriented SBC activities, on the fish purchasing and consumption practices of rural, inland households. Findings from this study are urgently needed by small island developing states in order to make policy and investment decisions on how best to improve households' diets using locally available, nutrient-dense foods such as fish. Investments such as these are needed to break the cycle of malnutrition.

ELIGIBILITY:
Inclusion Criteria:

* The individual's household is situated in a village included in the study, within a 30km radius of a coastal treatment site.

Exclusion Criteria:

* The individual's household is not situated in a village included in the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 720 (Actual)
Dates: Start 2021-05-15 (Actual); Primary Completion 2021-09-19 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Per capita household fish consumption | 1 year
  measured as total quantity (g) of fish consumed by the household in the previous seven days divided by the number adult equivalents in the household.
Frequency of fish consumed at household level | 1 year
  measured as the number of days fish were consumed out of the previous seven days.

SECONDARY OUTCOMES:
Frequency of fish consumption in women | 1 year
  measured as the number of days fish were consumed out of the previous seven days.
Frequency of fish consumption in children | 1 year
  measured as the number of days fish were consumed out of the previous seven days.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Tilley, PhD, Principal Investigator — WorldFish
Locations (1):
- WorldFish Timor-Leste, Dili, Timor-Leste

IPD SHARING:
Plan to Share IPD: No
All data will be kept confidential. Data will be submitted daily via 3G for review by in-country researchers and only stored on password protected mobile phone tablets and laptops temporarily. Participants will be assigned randomly-generated ID numbers, and names and identifying information will be de-linked from the dataset. Data will be analysed for groups and no individual response will be identifiable. Survey data will be archived and accessible to only the research team and those approved by the entire research team. Anonymised datasets will be securely maintained indefinitely to facilitate future research for example pooled analysis with other studies for purposes of meta-analysis or multi-site analysis.

REFERENCES:
- [Derived] Tilley A, Byrd KA, Pincus L, Klumpyan K, Dobson K, Dos Reis Lopes J, Shikuku KM. A randomised controlled trial to test the effects of fish aggregating devices (FADs) and SBC activities promoting fish consumption in Timor-Leste: A study protocol. PLoS One. 2022 Jul 8;17(7):e0269221. doi: 10.1371/journal.pone.0269221. eCollection 2022. PMID 35802640